CLINICAL TRIAL: NCT03090061
Title: Reliability of Light Induced Fluorescence Intraoral Camera Versus Visual-Tactile Method in Assessment of Marginal Integrity of Resin Composite Restorations: Diagnostic Invivo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Adly, internal resident, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CEBC-CU-2017-03-14
Record Dates: First submitted 2017-03-13; First posted 2017-03-24 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Microleakage Around Resin Composite Restorations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will not be blind about the type of intervention/control assessment methods. However it will not be allowed amongst the examiners to exchange any information throughout the entire study period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light induced fluorescence intraoral camera (Experimental)
  Interventions: Diagnostic Test: Light induced fluorescence intraoral camera
- Visual-tactile assessment method according to FDI criteria (Active Comparator)
  Interventions: Diagnostic Test: Visual-tactile assessment method according to FDI criteria

INTERVENTIONS:
Diagnostic Test: Light induced fluorescence intraoral camera — assessment of marginal integrity of resin composite restorations by light induced fluorescence intraoral camera
  Arms: Light induced fluorescence intraoral camera
Diagnostic Test: Visual-tactile assessment method according to FDI criteria — assessment of marginal integrity of resin composite restorations by visual-tactile method that includes the use of mirror, FDI probe under good illumination condition,
  Arms: Visual-tactile assessment method according to FDI criteria

SUMMARY:
This study will be conducted to assess diagnostic predictive values of a light induced fluorescence intraoral camera versus those of the visual-tactile assessment method according to FDI criteria in clinical evaluation the margins of resin composite restorations

DETAILED DESCRIPTION:
Each patient should have at least one resin composite restoration. The restoration will be evaluated by two diagnostic methods.

Each examiner will record the dental findings using both the visual- tactile assessment method and the fluorescent-aided identification method. The visual-tactile assessment method includes the use of mirror, FDI probe under good illumination condition, while the fluorescent-aided identification method will be performed by light induced fluorescence intraoral camera then the reliability of each diagnostic tool will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be over 18 years of age.
* Patients should have an acceptable oral hygiene level.
* Patients must have at least one posterior resin composite restoration.

Exclusion Criteria:

* Patients with a compromised medical history.
* Severe or active periodontal disease.
* Heavy bruxism or a traumatic occlusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Repeatability for both diagnostic methods | 20 minutes
  Three examiners will record the dental findings of 29 resin composte restorations using both the intervention and control assessment methods. Each method will be repeated twice to calculate the repeatability. The intra-operator agreement will be evaluated using the kappa statistics.
Reproducibility for both diagnostic methods | 1 week
  Three examiners will record the dental findings of 29 resin composite restorations using both the intervention and control assessment methods. Each method will be repeated after one week interval to calculate the reproducibility. The inter-operator agreement will be evaluated using the kappa statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided